CLINICAL TRIAL: NCT05966168
Title: Tracking of Mechanically Sensed Atrial Activity During Exercise Using a Leadless Transcatheter Pacing System
Brief Title: Micra AV Tracking During Exercise Testing
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00112840
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Heart Block AV
Keywords: AV Heart Block; High-grade Heart Block; MICRA AV; Medtronic
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Micra AV Exercise Testing (Experimental): All participants will have Micra AV 2.0 implanted then undergo exercise testing while wearing Holter Monitor
  Interventions: Device: Medtronic Micra AV Device

INTERVENTIONS:
Device: Medtronic Micra AV Device — Participants will already be planned to have a Micra AV 2.0 device implanted. Participants will then undergo treadmill exercise testing and wear a Holter monitor to determine the effectiveness of the Micra AV 2.0 device during exercise or elevated heart rates.
  Other Names: Micra AV Tracking During Exercise

SUMMARY:
The purpose of this study is to determine the effectiveness of the Micra AV 2.0 device during exercise or elevated heart rates. Participation in research studies is voluntary. In this study, participants will already be planned to have a Micra AV 2.0 device implanted. Participants will then undergo treadmill exercise testing and wear a Holter monitor. For each participant, the tracking performance of the Micra AV 2.0 will be evaluated at rest and during exercise. Follow up visits will occur as part of standard of care and each participant will be enrolled in the study for up to 6 months.

DETAILED DESCRIPTION:
Participants will be screened and eligible participants who express informed consent will complete exercise testing and holter monitoring. For each participant, the tracking performance of the atrial mechanically sensed, ventricular pacing device will be assessed at rest and during exercise using exercise testing. For each test, the sinus rate trend will be recorded alongside the presence or absence of a mechanically sensed ventricular paced event (AM-VP) for each sinus beat. The average tracking index in each phase of exercise testing - rest, exercise, and recovery - and across the spectrum of achieved heart rates across the cohort will be calculated and reported. Holter monitoring will also be used to assess tracking index across the spectrum of heart rates achieved during routine daily activities across a 24 hour period.

After enrollment, the following baseline information will be assimilated from the medical record and will be collected if not already done based on routine clinical care: date of pacemaker implant, pacemaker implant location (high septum, mid septum, apex), cardiac disease history, and programmed pacemaker parameters.

Exercise testing will be performed between one week and six months after Micra AV implant. Participants will complete preparation for exercise testing according to institutional standards. Participants will be given instructions to take all prescribed medications, including antiarrhythmic drugs and AV nodal blocking agents, according to their usual schedule, including on the day of the test.

Participants will be provided with a holter monitor. Participants will begin wearing the monitor during the rest period at the start of the exercise testing protocol. Exercise testing will be completed using standardized Micra AV device programming settings: VDD mode with nominal maximal tracking rate. Auto programming will be used to initialize device parameter selection. Following completion of auto programming, a MAM test will be performed to assess atrial signal discrimination. A fixed A3 discrimination threshold will then be selected which is approximately 1.0 m/s2 greater than the isolated accelerometer A3 signal.10 Other sensing parameters will be adjusted as clinically indicated to optimize atrial signal discrimination. Each participant will undergo device monitoring accompanied by external telemetry for 20 minutes at rest, followed by a fitness level-appropriate standardized stress protocol (e.g., Bruce protocol, Naughton protocol, Eckland protocol) on the treadmill or recumbent bicycle. They will perform graded exercise until achieving a heart rate of 130 bpm, or until physical fatigue, limiting chest pain (or discomfort), marked ischemia, or a drop in blood pressure occur (if such symptoms develop prior to reaching the target heart rate), supervised by a clinician experienced in performing cardiac stress testing. Once reaching 130 bpm, participants will remain at the current stage on their exercise protocol until physical fatigue, limiting chest pain (or discomfort), marked ischemia, or a drop in blood pressure occurs, or up to a maximum of twenty total minutes of exercise. Participants will be asked to report level of perceived exertion and fatigue level at pre-determined intervals. Cardiac rhythm will be recorded using 12-lead telemetry throughout the rest, exercise, and recovery periods. If the tracking index during exercise is lower than 70%, atrial sensing will be optimized using a MAM test.

The following data will be collected during exercise testing: exercise protocol utilized, protocol stage achieved, baseline cardiac rhythm, characterization of atrial and/or ventricular tachyarrhythmias, resting heart rate, peak heart rate, peak blood pressure, perceived level of exertion and fatigue, total exercise time, total metabolic equivalents (METs) achieved, and reason for termination.

The following data will be abstracted from device interrogation and 12-lead telemetry following the test: total number of sinus atrial beats, total number of premature atrial complexes (PAC), total number of premature ventricular complexes (PVC), number of tracked events, number of non-tracked ventricular paced events, and number of ventricular beats resulting from native AV conduction. Participants will continue to wear the provided holter monitor for the remainder of the 24 hour period. The following data will be collected during holter monitoring: average heart rate, peak heart rate, minimum heart rate, characterization of atrial and/or ventricular tachyarrhythmias, total number of sinus atrial beats, total number of premature atrial complexes (PAC), total number of premature ventricular complexes (PVC), number of tracked events, number of non-tracked ventricular paced events, and number of ventricular beats resulting from native AV conduction. Patient charts will be reviewed at the time of study completion to report clinical outcomes including death, device extraction, and/or transition to a transvenous pacing system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Written informed consent
* Presence of a Micra AV leadless pacemaker with the Micra AV 2.0 algorithm and at least 50% RV pacing
* High grade atrioventricular heart block as the primary indication for permanent pacing
* Sinus rhythm
* Physical ability to walk on a treadmill or ride a recumbent bicycle for exercise testing

Exclusion Criteria:

* Earlier version of the Micra leadless pacemaker
* Intact atrioventricular conduction
* Persistent atrial fibrillation
* Those with absolute contraindications to exercise testing:
* Acute myocardial infarction (MI) within 2 days
* Ongoing unstable angina
* Uncontrolled cardiac arrhythmia with hemodynamic compromise
* Active endocarditis
* Symptomatic severe aortic stenosis
* Decompensated heart failure
* Acute pulmonary embolism, pulmonary infarction, or deep vein thrombosis
* Acute myocarditis or pericarditis
* Acute aortic dissection
* Physical disability that precludes safe and adequate testing
* Inability to consent
* Patient refusal to participate
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Average tracking index at rest | 6 months
  Calculated as the percentage of atrial mechanically sensed, ventricular paced event (AM-VP) divided by total VP percentage.
Average tracking index during exercise | 6 months
  Calculated as the percentage of atrial mechanically sensed, ventricular paced event (AM-VP) divided by total VP percentage.
Average tracking index during recovery | 6 months
  Calculated as the percentage of atrial mechanically sensed, ventricular paced event (AM-VP) divided by total VP percentage.

SECONDARY OUTCOMES:
Average total AV synchrony at rest | 6 months
  Calculated as AM-VP percentage plus AM-VS percentage.
Average total AV synchrony during exercise | 6 months
  Calculated as AM-VP percentage plus AM-VS percentage.
Average total AV synchrony during recovery | 6 months
  Calculated as AM-VP percentage plus AM-VS percentage.
Average tracking index | 6 months
  The average tracking index across the spectrum of achieved heart rates across the cohort, categorized in 10-bpm ranges, from 55 bpm to 135 bpm.
Average total AV synchrony | 6 months
  The average total AV synchrony across the spectrum of achieved heart rates across the cohort, categorized in 10-bpm ranges, from 55 bpm to 135 bpm.
Device programming features among those with tracking index >70% | 6 months
  Percent of patients using auto threshold and window modes, and average A3 window, A3 threshold, A4 window, and A4 threshold values.
Clinical and device features which differentiate those with low tracking index | 6 months
  Clinical and device features which differentiate those with low tracking index (<70% tracking with ≥20% ventricular pacing) during the initial exercise test from those with high tracking index (if such a subset of patients exists).
Average tracking index during holter monitoring | 6 months
  • Average tracking index during holter monitoring across the spectrum of achieved heart rates across the cohort, categorized in 10-bpm ranges, from 55 bpm to 135 bpm.
Timeframe of optimal programing | 6 months
  Time (minutes) required to optimize programming prior to exercise testing.

CONTACTS AND LOCATIONS:
Overall Officials: Camille Frazier-Mills, Principal Investigator — Duke Medicine - Cardiology
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No